CLINICAL TRIAL: NCT05542914
Title: Integration of Electronic SBI(RT) Into an HIV Testing Program to Reduce Substance Use and HIV Risk Behavior Among MSM in Argentina
Brief Title: Electronic SBI(RT) for MSM in Argentina
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated by NIH on March 21, 2025 due to new guidelines.
Sponsor: Florida State University (Other)
Collaborators: Nexo Asociacion Civil (Unknown)
Responsible Party: Principal Investigator, Ivan Balan, Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002530
Record Dates: First submitted 2022-09-06; First posted 2022-09-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Substance Abuse; HIV
Keywords: SBIRT; HIV Prevention; MSM
MeSH Terms: conditions — Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-SBI (Experimental): Electronic Screening and Brief Intervention for substance use and HIV risk reduction
  Interventions: Behavioral: electronic screening and brief intervention.; Behavioral: Men's Health Project (MHP)
- Assessment Only (Active Comparator): These individuals complete only the screening instruments, no brief intervention
  Interventions: Behavioral: electronic screening and brief intervention.; Behavioral: Men's Health Project (MHP)

INTERVENTIONS:
Behavioral: electronic screening and brief intervention. — e-SBIs is an evidence based approach to engage non-treatment-seeking individuals who use substances to reduce use or enter treatment. It consists of completing screening instruments related to substance use and sexual risk behavior and receiving a tablet-based, Motivational Interviewing intervention to help individuals build motivation to reduce their use and plans to achieve their substance use and HIV risk reduction goals.
Behavioral: Men's Health Project (MHP) — This intervention will be offered to participants with moderate or greater severity substance use. This is a 4-session Motivational interviewing based intervention that has shown efficacy in prior studies. We are providing this as a possible referral program for study participants (either arm) who are interested in receiving substance abuse intervention.

SUMMARY:
Men who have sex with men (MSM) are disproportionally affected by HIV and substance abuse in the U.S., Europe, and Latin America. However, as in the general population, identifying and engaging MSM with problematic substance use (PSU) into treatment is a significant challenge, which results in the great majority of MSM with PSU never receiving treatment. The proposed study seeks to develop and pilot an electronic-Screening, Brief Intervention, Referral to Treatment (e-SBI-RT)program tailored for MSM awaiting their HIV test at Nexo Asociacion Civil, our community partners in Buenos Aires. The tablet-based e-SBI will integrate substance use and sexual risk behavior screeners and individually tailored Motivational Interviewing (MI) as the BI. We will also adapt and pilot the implementation of the Young Men's Health Project (from YMHP to MHP) a four-session MI-based intervention that effectively reduced substance use and condomless anal intercourse among substance using MSM. The Specific Aims of this R34 study are to: 1) develop the e-SBI intervention for MSM in an HIV testing context to reduce substance use and HIV risk behavior (Primary); 2) assess the feasibility and acceptability of integrating e-SBI into the HIV testing process at Nexo; and 3) assess the feasibility and acceptability of implementing adapted YMHP at Nexo. In Stage 1 (Development) we will develop e-SBI, adapt YMHP into MHP, train MHP counselors, and pilot e-SBI with 50 MSM coming to Nexo for HIV testing. In Stage 2 (RCT Pilot), we will randomize 200 MSM coming to Nexo for HIV testing at a 3:1 ratio (eSBI: Screening Assessments Only-SA) to assess the feasibility and acceptability of e-SBI among MSM coming to Nexo for HIV testing and establish and pilot the RCT process for a future trial. As a secondary aim, we will assess uptake, acceptability, and feasibility of delivering MHP to participants with low or moderate risk substance use and subsequent referrals to substance abuse treatment among participants with high-risk substance use or dependence. Lastly, we will explore preliminary findings on substance use and sexual risk reduction outcomes.

DETAILED DESCRIPTION:
This proposed study consists of two stages. Stage 1: Development will consist of developing e-SBI, the adaptation of YMHP into MHP, training counselors to deliver MHP, and piloting e-SBI with 50 MSM coming to Nexo for HIV testing. During the Stage 2: RCT Pilot, we will randomize 200 MSM coming to Nexo for HIV testing at a 3:1 ratio (eSBI: Screening Assessments Only-SA) to assess the feasibility and acceptability of e-SBI among MSM coming to Nexo for HIV testing and establish and pilot the RCT process for a future trial. As a secondary aim, we will assess uptake, acceptability, and feasibility of delivering MHP to participants with moderate risk substance use and subsequent referrals to SATx among participants with high-risk substance use or dependence. Lastly, we will explore preliminary findings on substance use and sexual risk reduction outcomes.

3.3.4. Stage 1: Development. 3.3.4.1. Development of e-SBI. Development of e-SBI app will be guided by the User Centered Rapid Application Development process (UCRAD). UCRAD merges the streamlined, iterative Rapid Application Development (RAD) approach with the User Centered Design approach (UC) which engages intended users throughout the app development process. This integrated approach aims to develop successful apps with good functionality, simple features, and a usable interface. As such, intended users are given access to prototypes of the app, allowing them to provide feedback before the next iteration of the app. UCRAD uses a three-phase process, as follows: Pre-design and interface prototyping, System architecture and coding, Deployment.

3.3.4.1.A Pre-design and interface prototyping. To accomplish this phase of UCRAD will obtain feedback from the Community Advisory Board regarding the study screening instruments (see below) and preliminary plans for the e-SBI content. After incorporating their feedback, we will conduct two focus groups (FGs) with MSM (N=16) recruited from Nexo testing clients who are 18+ years of age. They will complete a substance use screener consisting of the Illicit drug use question on the NIDA-modified ASSIST brief screen and the AUDIT-C (a 3-item alcohol use screen). Those who indicate using illicit drugs at least monthly and/or receive a score ≥4 on the AUDIT C will be eligible to participate. After completing informed consent, they will each complete paper and pencil versions of the screening instruments planned for inclusion in e-SBI. The 90-minute audio-recorded FGs will: 1) explore participants' reaction to the screeners and their impact on risk perception and motivation to reduce PSU and risk behavior; 2) evoke content for the BI component to develop menus of options for reasons to change and potential approaches to reduce problem substance use (PSU) and sexual risk behavior from which e-SBI users can choose. Within 48 hours of completing the FG, we will initiate a rapid analysis of this data using a qualitative matrix onto which participants responses and recommendations will be entered to quickly organize and summarize FG findings. These findings will be used to build the prototype of the e-SBI.

3.3.4.1.B System architecture and coding. This Phase 2 iterative app development process will be conducted with waves of 6 MSM also recruited from Nexo testing clients, with the same inclusion criteria as in the FGs. They will be recruited during two-week intervals to maintain a steady pace of feedback and revisions. Participants will complete the intervention on the tablet. Then, they will complete a 7-item self-report acceptability assessment. Afterwards, participants will be debriefed during an audio-recorded interview to explore four main areas: 1) their responses to the acceptability assessment; 2) overall reactions to e-SBI; 3) emotional reactions as e-SBI progressed, including heightened risk awareness, concern, or motivation to reduce substance use and sexual risk behavior; and 4) recommendations for improving the ability of the e-SBI to engage MSM who high-risk drugs and/or alcohol use into treatment. Interview data will undergo the same matrix-based, rapid analysis process used for the FG to quickly inform the next revision of the intervention. This process will be repeated with waves of 6 participants until mean scores on each acceptability question are ≥4.0 (≤2.0 on annoying), which we expect within 3-4 cycles. Development of the e-SBI will be guided by Choice Theory which has been used extensively to inform goal choice interventions, including MI interventions to reduce substance use among MSM. Rather than pre-set outcome expectations (ie., abstinence), goal choice interventions highlight personal choice and goal setting to engage individuals to reduce drug and alcohol use. Goal choice interventions appear to be equally effective as those that are abstinence-based and allowing individuals to set their own treatment goals appears to increase success rates.

3.3.4.1.C. Deployment. The initial version of the e-SBI will be deployed with 50 MSM coming to Nexo for HIV testing, to be used while they await their HIV test. After undergoing informed consent, these individuals will complete the eSBI, a brief quantitative acceptability assessment, and then proceed to have their HIV test (to minimize participant distress). Afterwards, up to 25 of these participants will be randomly selected (5 with low-risk substance use, 20 with moderate or high-risk substance use) to undergo an audio-recorded IDI. These IDIs will be guided by the Theoretical Framework of Acceptability (TFA) which was derived from a review of the literature on acceptability, and views acceptability as "a multi-faceted construct that reflects the extent to which people delivering or receiving a healthcare intervention consider it to be appropriate, based on anticipated or experienced cognitive and emotional responses to the intervention." These IDIs will be transcribed and uploaded to Dedoose for analysis. Additionally, we will use findings from these IDIs to finetune wording for a TFA-based quantitative assessments of acceptability that we will incorporate into the assessment battery during the Stage 2 RCT.

3.3.4.2. Adaptation of YMHP. MI interventions are used effectively globally including in Argentina, and MI and SBIRT have been effective with Latinos in the U.S. which suggests that YMHP may be easily tailored to the Argentine context. In consultation with our CAB, Dr. Balán, Lic. Marone, and Nexo counselors will adapt YMPH, guided by the modified ADAPT-ITT framework. The adaptation will focus on three main areas: 1) tailoring YMHP to Argentine MSM (including translation, cultural relevance for MSM over 29 years old); 2) we will adapt YMPH from a stand-alone intervention to an intervention within an SBIRT program by minimizing duplication with e-SBI content and incorporating content to improve linkage to specialized SATx for participants with high-risk substance use or dependence; and 3) adding content to address its poorer efficacy among partnered MSM. During this process, we will also train YMHP counselors in Motivational Interviewing and YMHP, with their skills assessed with the Motivational Interviewing Treatment Integrity V.4 (MITI-4) scale, which captures the counselor's level of fidelity to MI and establishes specific criteria for "Proficiency" in MI. Testing of the revised intervention will occur during the Stage 2, RCT pilot.

3.3.5. Stage 2: RCT Pilot We will assess feasibility and acceptability of e-SBI and conduct a preliminary exploration of substance use and sexual risk reduction outcomes. As a secondary aim, we will also assess uptake, acceptability, and feasibility of delivering MHP at Nexo and subsequent linkage to SATx among those with high-risk substance use or dependence.

3.3.5.1. Recruitment. MSM coming to Nexo for HIV testing and who are 18 years of age or older will be offered participation in the study. These clients will be given a flyer that, consistent with goal choice interventions, will create a low threshold for study participation by stressing personal choice, goal selection, and an intervention tailored specifically for MSM to figure out how to best reduce behavior that puts them at risk of HIV infection. Clients who wish to participate will complete informed consent, be randomized immediately, and given a tablet logged on to their respective study arm (and disposable headphones) to complete their study procedures. Research staff will record the number of clients who refuse participation.

3.3.5.2. Baseline Assessment. Participants in both conditions will complete a demographics questionnaire then a self-administered tablet-based 30-day Timeline Followback (TLFB) to track days of drug use, number of alcoholic drinks, and HIV risk behavior, defined as anal sex with: 1) an HIV positive partner who they were not sure had an undetectable viral load, or 2) a partner who had not tested HIV negative within the past three months). After completing their respective condition (described below) all participants will complete quantitative acceptability assessments based on the TFA

3.3.5.3. RCT Study Conditions. 3.3.5.3.A. Intervention group participants. After completing the baseline assessment, the tablet will immediately lead these participants to the e-SBI. The e-SBI branching logic will allow the intervention to be tailored based on factors such as participants' substance use risk level (based on ASSIST and AUDIT score), risk perception, and readiness to change. The e-SBI will also target the participant's sexual risk behavior and help them to develop a risk reduction plan, regardless of their substance use. Then, they will proceed to the usual HIV testing process at Nexo.

3.3.5.3.B. Control group participants. After completing the baseline assessment, the tablet will lead these participants to the same screening instruments as in the e-SBI but with no MI-based BI. Due to ethical considerations, control group participants with moderate or high-risk substance use based on the ASSIST or AUDIT scores will receive brief feedback on the tablet stating their level of risk, availability of MHP at Nexo, and instructions to see the receptionist for an appointment, if desired. Then, they will proceed to the usual HIV testing process at Nexo.

3.3.5.4. Referral for MHP. All individuals with moderate or high-risk substance use will be recommended for MHP (either actively motivated through e-SBI or informed about it in the control condition). MHP sessions will be conducted in-person at Nexo (later sessions can occur remotely, based on the participant's preference using a HIPAA compliant platform such as Zoom Healthcare). For participants with moderate risk substance use, MHP will focus on reducing substance use and sexual risk behavior. For participants with high-risk use or dependence, MHP sessions will focus on building motivation to enter specialized substance abuse treatment. To ensure intervention fidelity, all MHP sessions will be audio-recorded and rated using the MITI-4.

3.3.5.5. Follow-Up Assessments. All participants, including those who enter MHP or SATx, will repeat the self-administered 30-day TLFB at 3- and 6-months after enrollment to assess drug use, alcohol use, and sexual risk behavior. At 6-months they will also complete the screener instruments in the e-SBI, and TFA-based quantitative retrospective acceptability assessments of e-SBI and MHP (if they entered MHP), all of which will be programmed in RedCap and self-administered. We will also conduct IDIs with up to 45 participants (or less if saturation is reached), 15 with participants from either study condition who entered or completed MHP and/or SATx and 15 from each arm who met criteria for MHP but did not request it. These interviews will also guided by the TFA.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Stage 1 Focus Groups (FGs) and in-depth interviews (IDIs):

  1. Man who has had sex with men in the past 6 months;
  2. 18 years of age or older;
  3. Recently sought an HIV test at Nexo;
  4. Reports using drugs least once per month in the past 6 months and/or score 4 or greater on the AUDIT C, suggesting moderate risk alcohol use.

Participants in Stage 1 e-SBI pilot and the Stage 2 RCT:

1. Man who has had sex with men in the past 6 months
2. 18 years of age or older;
3. Currently seeking an HIV test at Nexo

Additional inclusion criteria for MHP entry:

1. Score of moderate or high risk drug or alcohol use based on the ASSIST and AUDIT, respectively

Exclusion Criteria:

* Exclusion Criteria for MHP entry:

  1. be in need of acute detoxification, as demonstrated by physical withdrawal symptoms or a history of withdrawal, such as previous delirium tremens or seizures
  2. reported regular use of opioids
  3. enrolled in concurrent drug- or alcohol-related treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as male or cis-gender male
Enrollment: 196 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate: Percent of MSM testing clients at Nexo who accept entry into the study | 8 months
  Will tabulate the percentage of MSM testing clients at Nexo who accept entry into the study vs those who refuse entry
Retention Rate: percent of participants who complete e-SBI | 6 months
  Will calculate the percent of participants who fully complete the e-SBI vs participants who do not complete the intervention
Mean overall acceptability rating of e-SBI from the TFA questionnaire | 6 months
  Will use the last question on the TFA questionnaire "Overall, how acceptable is the e-SBI to you?" to calculate mean overall acceptability and percent of participants who rate acceptability at 4 or higher.

SECONDARY OUTCOMES:
the percent of MSM with moderate or high-risk substance use who enter MHP from either RCT condition | 6 months
  We will assess the percent of MSM with moderate or high-risk alcohol and drug use based on the AUDIT and NIDA ASSIST who enter the MHP intervention
the percent of MHP participants who complete all four sessions | 6 months
  We will tabulate the number of sessions completed by each participant who enters MHP and identify the percent of MHP participants who complete all four intervention sessions
Mean overall acceptability rating of MHP from the TFA questionnaire | 6 months
  Will use the last question on the TFA questionnaire "Overall, how acceptable is MHP to you?" to calculate mean overall acceptability and percent of participants who rate acceptability at 4 or higher.
percentage of sessions conducted by each MHP counselor that meet criteria for MI proficiency | 6 months
  Will be assessed using the Motivational Interviewing Treatment Integrity (MITI.4) ratings.

OTHER OUTCOMES:
Occasions of drug use during the past month | 30 days
  Will use the 30-day Timeline Followback to assess
Occasions of heavy alcohol consumption (5+ drinks) during the past month | 30 days
  Will use the 30-day Timeline Followback to assess
Occasions of anal intercourse during the past month with a partner who is HIV positive or of unknown serostatus . | 30 days
  Will use the 30-day Timeline Followback to assess

CONTACTS AND LOCATIONS:
Overall Officials: Ivan C Balan, Principal Investigator — Florida State University, College of Medicine
Locations (1):
- Nexo Asociacion Civil, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
We will compile structured de-identified datasets and can make them available for additional/secondary data analyses. The research team will follow the "standards for privacy of individually identifiable health information." Participants' records and results will not be identified. No contact information will be included in any archived datasets. To preclude indirect identification, certain data elements such as date of birth will be transformed; date of birth will be used to provide a categorical age variable.
Time Frame: Starting 6 months after publication of main study findings.
Access Criteria: We will collaborate with and make our data available to other researchers for additional/secondary analyses. Dr. Balán and the research team will develop a process to review and approve data release based on concept sheets submitted by interested investigators and whether the data request is for new lines of analysis. Formal data sharing agreements will be developed to guide and encourage further data mining of the proposed datasets for various purposes

REFERENCES:
- [Derived] Balan IC, Marone RO, Barreda V, Naar S, Wang Y. Integration of an Electronic Screening, Brief Intervention, and Referral to Treatment Program Into an HIV Testing Program to Reduce Substance Use and HIV Risk Behavior Among Men Who Have Sex With Men: Protocol for Intervention Development and a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 14;13:e56683. doi: 10.2196/56683. PMID 38483463